CLINICAL TRIAL: NCT04258488
Title: Randomized, Evaluation of Long-term Anticoagulation With Oral Factor Xa Inhibitor Versus Vitamin K Antagonist After Mechanical Aortic Valve Replacement
Brief Title: Long-term Anticoagulation With Oral Factor Xa Inhibitor Versus Vitamin K Antagonist After Mechanical Aortic Valve Replacement
Acronym: RENOVATE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Joon Bum Kim (Other)
Responsible Party: Sponsor-Investigator, Joon Bum Kim, Professor, Department of Thoracic and Cardiovascular Surgery, University of Ulsan College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2020-01
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: AORTIC VALVE DISEASES; Thromboembolism
Keywords: Aortic valve replacement; Mechanical valve
MeSH Terms: conditions — Aortic Valve Disease; Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Factor Xa inhibitor (Experimental)
  Interventions: Drug: Rivaroxaban Oral Tablet
- Vitamin K antagonist (Active Comparator)
  Interventions: Drug: Vitamin K antagonist(warfarin)

INTERVENTIONS:
Drug: Rivaroxaban Oral Tablet — For 12months, Rivaroxaban oral tablet 20mg once daily For renal disorder subjects_creatinine clearance 15-49 mL/min, 15mg once daily
  Arms: Oral Factor Xa inhibitor
Drug: Vitamin K antagonist(warfarin) — For 12months, keep the international normalized ratio (INR) 1.7-3.0
  Arms: Vitamin K antagonist

SUMMARY:
This study evaluates the long-term anticoagulation with oral factor Xa inhibitor versus vitamin K antagonist in patients receiving a mechanical aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 and more
2. At least 3 months after mechanical aortic valve replacement
3. At least one of the conditions(as defined below) is met

   * The New York Heart Association (NYHA) Functional Classification I or II; or
   * According to the Valve Academic Research Consortium(VARC)2 criteria, confirmed proper valve function: no prosthesis-patient mismatch and mean aortic valve gradient <20 mm Hg or peak velocity <3 m/s, AND no moderate or severe prosthetic valve regurgitation
4. Voluntarily participated in the written agreement

Exclusion Criteria:

1. Old-generation mechanical valve
2. History of mechanical valve implantation in the mitral valve, pulmonary valve, or tricuspid valve
3. Valvular atrial fibrillation(atrial fibrillation with moderate or severe mitral stenosis)
4. Moderate to severe mitral stenosis or regurgitation
5. History of hemorrhagic stroke
6. Clinically overt stroke within the last 3 months
7. Renal failure(creatinine clearance <15mL/min) or on hemodialysis
8. Left ventricular dysfunction: Left ventricular ejection fraction (LVEF) ≤40%
9. Child-Pugh B and C hepatic impairment or any hepatic disease associated with coagulopathy
10. Clinically significant active bleeding
11. Bleeding or hemorrhagic disorder
12. The increased risk of bleeding due to the following reasons

    1. History of gastrointestinal ulcers or active ulcerations within the last 6 months
    2. History of intracranial or intracerebral hemorrhage within the last 6 months
    3. Spinal cord vascular abnormalities or intracerebral vascular abnormalities
    4. History of the brain, spinal cord, or ophthalmic surgery within the last 6 months
    5. History of the brain or spinal cord injury within the last 6 months
    6. History of the brain or spinal cord injury or spinal tap, major regional anesthesia, or spinal anesthesia within the last 6 months
    7. Esophageal varices
    8. Arteriovenous malformation
    9. Vascular aneurysms
    10. Malignant tumor with a high risk of bleeding
13. Bleeding tendencies associated with overt bleeding of

    1. gastrointestinal, genitourinary, respiratory tract, or colorectal cancer
    2. cerebrovascular hemorrhage
    3. aneurysms- cerebral, dissecting aorta
    4. pericarditis and pericardial effusions
    5. bacterial endocarditis
14. Hemodynamically unstable or pulmonary embolism required thrombolysis or embolectomy
15. Combination therapy with other anticoagulants(Unfractionated heparin(UFH), enoxaparin, dalteparin, fondaparinux, etc.) However, the following cases are permitted

    * Switching anticoagulants
    * Intravenous UFH to keep central/arterial lines open
16. Uncontrolled moderate or severe hypertension
17. Anemia at least one among the conditions(as defined below) is met 1) Hemoglobin level <10.0 g/dL or platelet count < 100 x 10x9/L within the last 6 months 2) Diagnosed and documented ongoing anemia
18. Infective endocarditis
19. Hypersensitivity to the main component or constituents of Rivaroxaban or Vitamin K antagonist
20. Positive pregnancy test results (all pregnant women should undergo urinary human chorionic gonadotropin (hCG) testing within 7 days before screening and/or randomization) or during pregnancy or lactation
21. A genetic problem with galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
22. The unsuitable condition of the protocol
23. Actively participating in another drug or device investigational study, which has not completed the primary endpoint follow-up period
24. Terminal illness with life expectancy <12 months
25. Vitamin K deficiency
26. Alcoholic or psychical disorder
27. Threatened abortion, eclampsia, or preeclampsia
28. Concomitant use with antiplatelet in patients with a history of stroke or transient ischemic attack for the treatment of the acute coronary syndrome

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with the composite of cardiac death, valve thrombosis, valve-related thromboembolic event, major bleeding, and clinically-relevant non-major bleeding | 1 year
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event that is considered to have occurred if any one of several different events is observed.
  Clinically-relevant non-major bleeding is defined as BARC(Bleeding Academic Research Consortium) 2 Bleeding and major Bleeding is defined as BARC(Bleeding Academic Research Consortium) 3 or 5 Bleeding.

SECONDARY OUTCOMES:
Number of Participants With all cause death | 1 year
Number of Participants With cardiovascular death | 1 year
Number of Participants With valve thrombosis confirmed by transthoracic echocardiography, transesophageal echocardiography, cine fluoroscopy, computed tomography, or autopsy (Valve Academic Research Consortium (VARC ) criteria) | 1 year
Number of Participants With valve-related thromboembolic | 1 year
Number of Participants With transient ischemic attack | 1 year
Number of Participants With stroke | 1 year
Number of Participants With systemic embolism | 1 year
Number of Participants With myocardial infarction | 1 year
Number of Participants With major bleeding | 1 year
  BARC (Bleeding Academic Research Consortium) 3 or 5
Number of Participants With Clinically-relevant non-major bleeding | 1 year
  BARC (Bleeding Academic Research Consortium) 2
Number of Participants With the composite of cardiac death, valve thrombosis and valve-related thromboembolic event | 1 year
Number of Participants With the composite of cardiac death, valve thrombosis, stroke, systemic embolism and myocardial infarction event | 1 year
Number of Participants With the composite event of major bleeding and clinically-relevant non-major bleeding | 1 year
  Clinically-relevant non-major bleeding is defined as BARC (Bleeding Academic Research Consortium) 2 Bleeding and major Bleeding is defined as BARC (Bleeding Academic Research Consortium) 3 or 5 Bleeding.
Number of Participants With the composite of stroke, systemic embolism, transient ischemic attack and myocardial infarction event | 1 year
Number of Participants With the composite of all-cause death, stroke, systemic embolism, transient ischemic attack and myocardial infarction event | 1 year
The change of echocardiographic parameter | 1 year
  Integral ratio at baseline and 1 year follow-up : transaortic valve mean gradient
The change of echocardiographic parameter | 1 year
  Integral ratio at baseline and 1 year follow-up : transaortic valve peak gradient
The change of echocardiographic parameter | 1 year
  Integral ratio at baseline and 1 year follow-up : transaortic valve peak velocity
The change of echocardiographic parameter | 1 year
  Integral ratio at baseline and 1 year follow-up : effective orifice area(EOA)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-min Ahn, MD, Principal Investigator — drjmahn@gmail.com
Locations (15):
- South Korea (15):
  - Buchen Sejong Hospital, Bucheon-si
  - Seoul National University Bundang Hospital, Bundang
  - Dong-A University Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - GangNeung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon
  - St. Vincent's Hospital, Catholic University of Korea, Suwon
  - Eulji University Uijeongbu Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: Undecided